CLINICAL TRIAL: NCT00040053
Title: Double-Blind, Placebo-Controlled, Dose Response Trial of Ondansetron for the Treatment of Methamphetamine Dependence.
Brief Title: Ondansetron for the Treatment of Methamphetamine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0011-1
Record Dates: First submitted 2002-06-18; First posted 2002-06-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Amphetamine-Related Disorders
Keywords: amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Ondansetron

INTERVENTIONS:
Drug: Ondansetron

SUMMARY:
The purpose of this study is to assess ondansetron for the treatment of methamphetamine dependence.

DETAILED DESCRIPTION:
This study was designed to be a preliminary assessment of the efficacy and safety of 3-wide range doses of ondansetron (0.25, 1.0 and 4.0 mg taken orally twice per day) to reduce methamphetamine use in subjects with methamphetamine dependence and to determine the optimal dose of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

18 years of age. Treatment seeking for meth dependence.

Exclusion Criteria:

Please contact site director for more details.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154
Dates: Start 2002-06; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Clinicial improvement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (6):
- United States (6):
  - South Bay Treatment Center, Chula Vista, California
  - Matrix Institute on Addictions, Costa Mesa, California
  - John A. Burns School of Medicine, Honolulu, Hawaii
  - Powell Chemical Dependency Center, Des Moines, Iowa
  - University of Missouri - Kansas City, Kansas City, Missouri
  - University of Texas Health Science Center, Houston, Texas